CLINICAL TRIAL: NCT01624077
Title: Phase 1 Clinical Trial Using Regulatory T Cells as Individualized Medicine to Promote Donor-specific Clinical Liver Transplantation Tolerance in Nanjing
Brief Title: Safety Study of Using Regulatory T Cells Induce Liver Transplantation Tolerance
Acronym: Treg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Ling Lu, Liver transplantation Center, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJLT001
Record Dates: First submitted 2012-01-16; First posted 2012-06-20 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Rejection of Liver Transplant
Keywords: Regulatory T cells; Liver Transplantation; Rejection; Tolerance; Cell tolerance; Survival
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regulatory T cells (Experimental): Naïve CD4+ T cells isolated from peripheral blood mononuclear cells were stimulated with GMP anti-CD3/CD28 coated beads in the presence of IL-2 ,TGF-β.
  Interventions: Biological: Regulatory T cells

INTERVENTIONS:
Biological: Regulatory T cells — Tregs will inject after liver transplantation
  Other Names: Treg

SUMMARY:
The first trial will involve the generation of donor alloantigen-specific CD4+CD25+ Tregs from peripheral blood of pre-transplant patients, the administration of the CD4+CD25+ Tregs (1 x 106 cells/kg) at several intervals (for graft specific tolerance induction).

DETAILED DESCRIPTION:
The first trial will involve the generation of CD4+CD25+CD127- Tregs from peripheral blood of pre-transplant patients, followed by a course (up to 24 months) of tacrolimus (5-10 ng/ml) treatment (to prevent chronic rejection) and the administration of the CD4+CD25+CD127- Tregs (1 x 106 cells/kg) at several intervals (for tolerance induction). The immunesuppress drugs will be gradully withdraw within one year. The number of CD4+CD25+ Tregs needed is based on the assumption that the frequencies of alloreactive CD4+ T cells with direct and indirect allospecificity were 1/104 and 1/105, respectively.

The second trial will be carried out in 1-10 year post living donor liver transplantation patients currently under immunosuppressive drug treatment. The investigators will isolate CD4+CD25+CD127- Tregs from these patients, and expand them with mismatched living donor antigens. The patients will be subsequently treated with the expanded donor-antigen specific CD4+CD25+CD127- Tregs (1 x 106 cells/kg) at several intervals, and immunosuppressive drug treatment will be withdrawn.

In both clinical trials, the investigators will monitor the number of allospecific Tregs in patients at different time periods, and to test their suppressive functions in vitro. If there will be any signs of graft rejection, patients will be switched back to immunosuppressive drug treatment. The investigators expect that the innovative Tregs immunosuppressive regimen will lead to achieve permanent liver transplantation tolerance without the use of conventional immunosuppressive drugs: the holygrail in clinical transplantation medicine.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than 50kg
* Will be receiving a living-related primary liver allograft
* Negative B-cell and T-cell cytotoxic and flow cytometry crossmatch
* Normal echocardiogram (ECG) with an ejection fraction of greater than 50%
* Parents willing to comply with the study visits

Exclusion Criteria:

* Current active infection
* Pregnant or breastfeeding
* Evidence of HIV infection or known HIV positive serology
* Antibody positive for hepatitis C virus
* Surface antigen positive for HBV
* Recipient or donor is positive for tuberculosis (TB), under treatment for suspected TB, or previously exposed to TB (positive Mantoux test)
* Current cancer or a history of cancer
* Uncontrolled concomitant infections, severe diarrhea, vomiting, active upper gastrointestinal tract malabsorption, active peptic ulcer, or any other unstable medical condition that could interfere with this study
* Currently receiving an investigational drug or received an investigational drug within 30 days prior to transplant
* Currently receiving any immunosuppressive agent
* Anticipated contraindication to taking medications orally or via nasogastric tube by the morning of Day 2 following completion of the transplant procedure
* Require certain medications
* Known hypersensitivity to any of the study medications,
* Any form of substance abuse, psychiatric disorder, or other condition that, in opinion of the investigator, may interfere with the study
* Anticipated contraindication to study medications administration for longer than 5 days post-transplant
* History of rejection after organ transplantation
* Muti-organ transplantation
* Autoimmune disease

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Patient and graft survival | one year posttransplantation

SECONDARY OUTCOMES:
Patient and graft survival | 3 years post transplantation
Incidence rate of biopsy-proven acute or chronic organ rejection | 3 years post transplantation
Incidence of adverse events associated with liver transplantation and immunosuppression | 3 years posttransplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wang, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing Medical University, Nanjing, Jiangsu, China